CLINICAL TRIAL: NCT05925907
Title: Ciss-DLV-Cross-cultural Adaptation of the 'Cold Intolerance Severity Score' (CISS) to the Dutch Language.
Brief Title: Cross-cultural Adaptation of the 'Cold Intolerance Severity Score' (CISS) to the Dutch Language.
Acronym: Ciss-DLV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Handcentrum, Bilthoven, The Netherlands (Unknown)
Responsible Party: Principal Investigator, Reinier Feitz, MD PhD, Reinier Feitz, MD, PhD, plastic surgeon, Erasmus Medical Center
Other Study IDs: PANAMA-10267
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Hand Injuries
Keywords: CISS, handsurgery, crush, nerve injury , amputation, coldintolerance
MeSH Terms: conditions — Hand Injuries; Crisponi syndrome; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Handsurgery patients: patients recruited from trauma handsurgery outpatient clinic in an academic teaching hospital, level 1 trauma unit.
- Medicolegal patients: Medicolegal patients that are examined in order to asses their personal injury claim.

SUMMARY:
To report Cold intolerance by the CISS score in medicolegal patients.

DETAILED DESCRIPTION:
Rationale Cold intolerance is an important finding in hand trauma patients, nerve injury, crush injury, degloving injury or amputation. Cold intolerance as a symptom is probably the least responsive to any known medical treatment.

Perhaps due to the fact that we have no control over it, the consequences for cold tolerance are seldom researched. patients involved in medicolegal claims report more pain and less function than controls. Medicolegal examinations for various indications offer a long-term outcome view for the symptoms of cold tolerance. Therefore, together with Handcentrum we want to translate, improve and test the current PROM for cold intolerance CISS

Objective To report Coldintolerance by the CISS score in medicolegal patients.

Study parameters / Endpoints A validated Dutch version of the CISS A report on 100 CISS scores in medicolegal patients Examine if a shorter version of the CISS questionnaire is feasible

Study design 2-3 independent forward translations (e.g. from English into Dutch) by native speakers of the target language (e.g. Dutch). One of the translators understands the concept, one translator has no knowledge of the concept that the questionnaire measures and no medical background.

The translators make a joint forward translation together with an independent person.

2-3 independent back-translations (e.g. from Dutch into English) by native speakers of the source language (e.g. English). Both translators have no knowledge of the concept the questionnaire measures and have no medical background. ... Read more

Burden and risk These questionnaires are mandatory anyway. So, no additional time for the patients needed. There is no risk involved. There is no alteration in the medical or clinical pathway.

Recruitment and consent automatically enrolment and permission via Medisoft software from HandC

Summary Translation and validation of a Dutch version of a PROM for cold intolerance

ELIGIBILITY:
Inclusion Criteria:

* - Adult
* Traumatic hand injury
* Sufficient knowledge of the Dutch language (at least level B1)

Exclusion Criteria:

* - Definitive total hand amputation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Handsurgery patients and medicolegal patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Validation of a Dutch language translation of standard cold intolerance form | 1 year
  Test and retest of a Dutch language model of the CISS score

CONTACTS AND LOCATIONS:
Overall Officials: Reinier Feitz, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmuc MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided